CLINICAL TRIAL: NCT01269723
Title: Effects of Sulforaphane (SFN)on Innate Immune Responses to Live Attenuated Influenza Virus in Smokers and Nonsmokers
Brief Title: Effects of Sulforaphane (SFN) on Immune Response to Live Attenuated Influenza Virus in Smokers and Nonsmokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Terry Noah, MD, Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 10-1806; R01HL095163-02 (NIH)
Record Dates: First submitted 2010-12-14; First posted 2011-01-04 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Smoking
Keywords: Smoking; influenza; influenza vaccine
MeSH Terms: conditions — Smoking; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Broccoli sprout homogenate (Active Comparator): The broccoli sprouts and water are chopped in a blender until a uniform mix is obtained. Salt or sugar may be added to the "shake".
  Interventions: Dietary Supplement: Broccoli sprout homogenate
- alfalfa sprout homogenate (Placebo Comparator): Alfalfa sprouts and water are chopped in a blender until a uniform mix is obtained. Salt or sugar may be added to the "shake".
  Interventions: Dietary Supplement: Alfalfa sprout homogenate

INTERVENTIONS:
Dietary Supplement: Broccoli sprout homogenate — Subjects will drink the broccoli shake homogenate
  Other Names: Broccoli sprout shake
  Arms: Broccoli sprout homogenate
Dietary Supplement: Alfalfa sprout homogenate — Subjects will drink the alfalfa sprout homogenate.
  Other Names: Alfalfa sprout shake
  Arms: alfalfa sprout homogenate

SUMMARY:
Vegetables such as broccoli, cauliflower, kale and cabbage are particularly rich in a plant chemical called sulforaphane (SFN) which boosts production of certain "defense" enzymes that increase the activity of antioxidants. In animals, the chemical protection from SFN helps prevent diseases associated with inflammation and cancer among others, and this is currently being studied in humans.

Young broccoli sprouts have a particularly high level of SFN compared to other foods. The purpose of this research study is to learn about short term responses to live attenuated influenza virus (LAIV, administered to you via Flumist® vaccine) between smoking and nonsmoking volunteers treated with broccoli sprout homogenates ("shake") or a placebo homogenate. This will be done by obtaining a series of "nasal lavages" or rinses of your nose with salt water, as well as 3 superficial biopsies of the inside lining of your nose both before and after you receive the vaccine. Using these samples, we will measure the amount of virus and the amount of inflammation in your nose and compare how smokers and nonsmokers respond to the vaccine when they are given a broccoli sprout homogenate (high in SFN) or a placebo alfalfa spout "shake" which is low in SFN during each of 4 study visits.

Subjects will be seen for a screening visit (inc. HIV test) and then randomly assigned to receive 1 of 2 homogenates. Broccoli sprout homogenate will be the the active treatment arm while the placebo arm will be alfalfa sprout homogenate. Two to 4 weeks after screening, subjects will return for 5 sequential visits (Monday-Friday). Monday-Thursday they will receive the assigned homogenate. On Tuesday, they will receive the Flumist®vaccine. Subjects will also be seen at 1 and 3 weeks post vaccine. Nasal lavage (NL), blood samples and nasal biopsies will performed prior to and after study interventions.

DETAILED DESCRIPTION:
Schedule of visits:

Prior to the screening visit, subjects will be asked to avoid cruciferous vegetables (list will be provided to them), corticosteroids and nonsteroidal anti-inflammatory medications for 1 week prior to the initial visit and again for 1 week prior to all remaining visits. They will to also be asked to avoid antioxidant vitamins as well as juices/drinks with added vitamin supplements for 2 days prior to enrollment through study completion.

Baseline screening: obtain informed consent, review medical history, concomitant medications, vital signs (VS's), urine collection for analysis of cotinine and SFN metabolites for all subjects and urine pregnancy test for females of child bearing potential (all female subjects unless they are s/p oophorectomy), physical exam by study MD, complete symptom scoring, collect nasal lavage, and nasal biopsy (both nares), buccal swab collection and venipuncture (up to 75 cc's) will be performed for human immunodeficiency virus (HIV) test, baseline SFN level, immune mediators and SFN-induced gene expression changes. Food diaries will be provided with instructions for subjects at this visit

After successful completion of the screening, the subject will be randomized to receive broccoli sprout homogenates or alfalfa sprout homogenates during the next 4 study visits. Subjects will return 2-4 weeks after screening for 5 daily sequential visits (Monday through Friday).

Monday (Day -1): VS's, review of concomitant medications, urine collection for analysis of cotinine and SFN metabolites for all subjects and Hcg for females of child bearing potential, nasal lavage, observed ingestion of initial dose and continue food diaries started 3 days prior.

Tuesday (Day 0): VS's, symptom/adverse event evaluation, review of concomitant medications, urine collection for analysis of cotinine and SFN metabolites, observed ingestion of 2nd dose, NL, administration of LAIV, continue food diaries.

Wednesday (Day 1): VS's, symptom/adverse event evaluation, review of concomitant medications, urine collection for analysis of cotinine and SFN metabolites, observed ingestion of 3rd dose, NL and continue food diaries.

Thursday (Day 2): VS's, symptom/adverse event evaluation, review of concomitant medications and observed ingestion of 4th dose. Two hours after ingestion, urine collection for analysis of cotinine and SFN metabolites, venipuncture (up to 10 cc's for SFN level), nasal biopsy (left nare) and NL will be performed. Continue food diaries.

Friday (Day 3): VS's, symptom/adverse event evaluation, review of concomitant medications, urine collection for analysis of cotinine and SFN metabolites, NL, continue food diaries.

Day 7 (+/- 1 day): VS's, symptom/adverse event evaluation, review of concomitant medications, urine collection for analysis of cotinine and SFN metabolites, nasal biopsy (right nare), NL, continue food diaries.

Day 21 (+/- 1 week): VS's, symptom/adverse event evaluation, review of concomitant medications urine collection for analysis of cotinine and SFN metabolites, NL, venipuncture (up to 45 cc's) for immune mediators as well as SFN-induced gene expression changes and anti-influenza antibody level, collect completed food diary

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, age 18-40 yr who are either nonsmokers OR smokers (> 0.5 pack/day);
* Willing to avoid corticosteroids and nonsteroidal anti-inflammatory medications for 1 week prior to study entry and again for 1 week prior to all remaining visits;
* Willing to avoid antioxidant vitamins and cruciferous vegetables as well as juices/drinks with vitamin supplements added for 2 days prior to Day (-1) of the protocol and throughout the subsequent study.

Exclusion Criteria:

* Symptomatic allergies requiring medications for at least a 2 week interval during the past year;
* Respiratory infection (cough, sore throat, sinusitis, fever etc) within prior 4 weeks;
* Current nutritional disorder such as anorexia, bulimia, irritable bowel syndrome, Crohn's disease etc;
* Pregnancy or nursing;
* Asthma (other than wheezing occurring only in childhood); immunodeficiency (HIV or other); or any chronic medical condition that, in the opinion of the investigator, would preclude subject participation;
* Current use of immunosuppressive drugs;
* History of fainting or feeling severely dizzy with blood draws;
* History of hypersensitivity, especially anaphylactic reactions, to egg proteins, gentamicin, gelatin, or arginine or with adverse reactions to previous influenza vaccinations;
* History of Guillain Barre syndrome;
* Smokers who have abnormal lung function on pulmonary function testing at the time of screening (FVC and FEV1 < 80% of that predicted based on subject age, gender, height and race);
* Subjects who will be unable to avoid contact with immunocompromised individuals for 3 weeks after receiving LAIV vaccine;
* Receipt of any type of influenza vaccine since August 2009;
* Diagnosed influenza illness since August 2009;
* History of intolerance of or aversion to broccoli.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 (IL-6) in NL after LAIV inoculation (expressed as area under curve for ratio of IL-6 to baseline) in smokers | at days 1, 2 ,3, 7 and 21 post LAIV
  This will be performed by repetitive spraying of sterile normal saline irrigation solution (5 ml total) into the nostril, followed by voluntary expelling of fluid by the subject into a specimen collection cup. Both nostrils are lavaged in this way and the resulting nasal lavage fluid (NLF) from both sides is combined.

SECONDARY OUTCOMES:
change in nasal cells-cytokines, chemokines, natural killer cell activation; tolerance of homogenate; nasal biopsy Nrf2, cytokine, and phase II enzyme mRNA; serum antibodies; blood cell response to influenza antigen | For nasal lavage-at days 1, 2 ,3, 7 and 21 post LAIV; for biopsy samples taken on Days 2 and 7 post LAIV; for blood endpoints-Days 2 and 21 post LAIV
  Nasal lavage is as previously described. Blood collection will be via venipuncture and nasal epithelial cells will be collected during a nasal scrape.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina at Chapel Hill School of Medicine
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Muller L, Meyer M, Bauer RN, Zhou H, Zhang H, Jones S, Robinette C, Noah TL, Jaspers I. Effect of Broccoli Sprouts and Live Attenuated Influenza Virus on Peripheral Blood Natural Killer Cells: A Randomized, Double-Blind Study. PLoS One. 2016 Jan 28;11(1):e0147742. doi: 10.1371/journal.pone.0147742. eCollection 2016. PMID 26820305
- [Derived] Noah TL, Zhang H, Zhou H, Glista-Baker E, Muller L, Bauer RN, Meyer M, Murphy PC, Jones S, Letang B, Robinette C, Jaspers I. Effect of broccoli sprouts on nasal response to live attenuated influenza virus in smokers: a randomized, double-blind study. PLoS One. 2014 Jun 9;9(6):e98671. doi: 10.1371/journal.pone.0098671. eCollection 2014. PMID 24910991